CLINICAL TRIAL: NCT00856336
Title: 5,6-Dimethylxanthenone-4-Acetic Acid (DMXAA) in the Treatment of Refractory Tumors: A Phase I Multicentre Doubleblind Randomized Six-Way Intrapatient Dose-Ranging Crossover Safety Study.
Brief Title: Phase I Safety Study of DMXAA in Refractory Tumors
Acronym: DART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Chief Medical Officer, Antisoma Research Limited
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DART
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Refractory Tumors
MeSH Terms: conditions — Neoplasms | interventions — vadimezan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: DMXAA — DMXAA, given intravenously over 20 minutes. Patients were to each undergo six doses of treatment at weekly intervals, receiving each of six doses (300, 600, 1200, 1800, 2400 and 3000 mg/m2)

SUMMARY:
This was a phase I study aimed at identifying safe doses of DMXAA (now known as ASA404) to be used in future combination studies with chemotherapy.

DETAILED DESCRIPTION:
This was a multi-centre randomized, double blind study to further characterize the effect of DMXAA on QTc interval, ophthalmic safety and pharmacodynamic effects on tumour blood flow.

Patients with refractory tumors were to each undergo six doses of treatment at weekly intervals, receiving each of six doses of DMXAA (300, 600, 1200, 1800, 2400 and 3000 mg/m2)

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of cancer, by histopathology or cytology, which was not amenable to any standard therapy or was refractory to conventional therapy
2. Age ≥ 18 years
3. Life expectancy of at least 12 weeks
4. WHO performance status of 0-2
5. Hematological and biochemical indices at the start of treatment:

   1. Hemoglobin at least 9 g/dl
   2. Leukocyte count at least 3.0 x 109/l
   3. Neutrophils at least 1.5 x 109/l
   4. Platelets at least 100 x 109/l
   5. Serum Creatinine not higher than140 μmol/l
   6. Liver function tests (ALT, AST, ALK PHOS) no higher than thrice the upper limit of the reference range, if no demonstrable liver metastases or no more than 5 x upper limit of the normal range in the presence of liver or bone metastases
   7. Absolute QTc interval values of less than 470 ms in females and less than 450 ms in males as assessed by the Investigator
6. Presence of a lesion which was amenable to dynamic MRI
7. Written informed consent and the ability of the patient to co-operate with treatment and follow up

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks prior to treatment
2. Pregnant or lactating women were excluded
3. Patients who were poor medical risks because of non-malignant systemic disease, as well as those with active uncontrolled infection
4. Current malignancies at other sites
5. Significant history of recreational drug abuse
6. Glucocorticosteroids in doses exceeding those required for physiological replacement within the previous 2 weeks
7. Skin lesions that may prevent long-term ECG acquisition
8. Body mass index above 30 kg/m2
9. Patients who were taking certain medications
10. Patients with clinical evidence of brain metastases
11. Patients with certain cardiac conditions

    1. Advancing or unstable ischemic heart disease
    2. Pacing devices and/or implantable cardiovertor-defibrillator
    3. Significant cardiovascular disease or any unstable cardiovascular disease
    4. Non-sustained or sustained atrial and/or ventricular tachyarrhythmias
    5. Atrial fibrillation (including paroxysmal atrial fibrillation) or atrial flutter
    6. Bundle Branch Block, any stable intra-cardiac conduction abnormality with QRS complex > 120 ms, any unstable intra-cardiac conduction abnormality
    7. Sick sinus syndrome, or sinus pauses > 2 seconds
    8. Known atrial and/or ventricular ectopic beats > 10/hour
    9. Fixed second degree AV block, transient or fixed third degree AV block
    10. History of documented ventricular flutter, ventricular fibrillation, Torsade de Pointes tachycardia
    11. Patients who had previously received anthracyclines or other known cardiotoxic medication
12. Women with breast implants as these may have interfered with the recording of the ECG
13. Patients with severe electrolyte abnormalities and patients in whom transient electrolyte abnormalities may have been expected during any visit of the study
14. Patients in whom concomitant neurotropic drug therapy was known to change or was likely to change during the course of the study, where such therapy was likely to affect the patients ERG measurement
15. Ophthalmic conditions where in the opinion of the investigator they might affect the recording of the ERG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-05; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
To identify a range of doses for DMXAA where there was either no effect or an acceptably small effect on QTc

SECONDARY OUTCOMES:
To investigate and describe the relationship between QTc prolongation, plasma levels of DMXAA and time from start of infusion.
To further investigate the safety profile of DMXAA
To further investigate the pharmacokinetic behaviour of DMXAA
To further characterise the ophthalmic effects of DMXAA
To document anti-tumour activity and/or clinical signs of efficacy in patients
To assess the effects of DMXAA on tumour blood flow using dynamic MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mark McKeage, Principal Investigator — The University of Auckland; Michael Jameson, Principal Investigator — Waikato Hospital; Mark Jeffery, Principal Investigator — Christchurch Hospital

REFERENCES:
- [Result] McKeage MJ, Fong P, Jeffery M, Baguley BC, Kestell P, Ravic M, Jameson MB. 5,6-Dimethylxanthenone-4-acetic acid in the treatment of refractory tumors: a phase I safety study of a vascular disrupting agent. Clin Cancer Res. 2006 Mar 15;12(6):1776-84. doi: 10.1158/1078-0432.CCR-05-1939. PMID 16551862
- [Derived] Jameson MB, Sharp DM, Sissingh JI, Hogg CR, Thompson PI, McKeage MJ, Jeffery M, Waller S, Acton G, Green C, Baguley BC. Transient retinal effects of 5,6-dimethylxanthenone-4-acetic acid (DMXAA, ASA404), an antitumor vascular-disrupting agent in phase I clinical trials. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2553-9. doi: 10.1167/iovs.08-2068. Epub 2009 Apr 22. PMID 19387077